CLINICAL TRIAL: NCT01165138
Title: HZA106827: A Randomised, Double-blind, Placebo-controlled (With Rescue Medication), Parallel Group Multicentre Study of Fluticasone Furoate/GW642444 Inhalation Powder and Fluticasone Furoate Inhalation Powder Alone in the Treatment of Persistent Asthma in Adults and Adolescents
Brief Title: Study HZA106827: Efficacy/Safety Study of Fluticasone Furoate/Vilanterol (GW642444) in Adult and Adolescent Asthmatics
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 106827
Record Dates: First submitted 2010-07-15; First posted 2010-07-19 (Estimated); Results first posted 2013-07-30 (Estimated); Last update posted 2018-02-14 (Actual); Status verified 2018-01

CONDITIONS: Asthma
Keywords: GW642444; Vilanterol; Asthma; Fluticasone Furoate
MeSH Terms: conditions — Asthma | interventions — fluticasone furoate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Fluticasone furoate/Vilanterol (GW642444) (Experimental): Fluticasone furoate/Vilanterol inhalation powder once daily for 12 weeks
  Interventions: Drug: Fluticasone furoate/Vilanterol Inhalation Powder
- Fluticasone Furoate (Experimental): Fluticasone furoate inhalation powder once daily for 12 weeks
  Interventions: Drug: Fluticasone Furoate Inhalation Powder
- Placebo (Placebo Comparator): Placebo inhalation powder once daily for 12 weeks
  Interventions: Drug: Placebo Inhaltion Powder

INTERVENTIONS:
Drug: Fluticasone furoate/Vilanterol Inhalation Powder — Fluticasone furoate/Vilanterol Inhalation Powder inhaled orally once daily for 12 weeks
  Arms: Fluticasone furoate/Vilanterol (GW642444)
Drug: Fluticasone Furoate Inhalation Powder — Fluticasone Furoate Inhalation Powder inhaled orally once daily for 12 weeks
  Arms: Fluticasone Furoate
Drug: Placebo Inhaltion Powder — Placebo Inhaltion Powder inhaled orally once daily for 12 weeks
  Arms: Placebo

SUMMARY:
The purpose of the study is to compare the efficacy and safety of fluticasone furoate/vilanterol (GW642444) inhalation powder and fluticasone furoate inhalation powder both administered once daily in adolescent and adult subjects 12 years of age and older with persistent bronchial asthma over a 12 week treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients at least 12 years of age
* Male and female; female subjects of childbearing potential must be willing to use birth control
* Pre-bronchodilator FEV1 of 40-90% predicted normal
* Reversibility FEV1 of at least 12% and 200mL
* Current asthma therapy includes inhaled corticosteroid use for at least 12 weeks prior to first visit

Exclusion Criteria:

* History of life-threatening asthma during last 10 years
* Respiratory infection or oral candidiasis
* Asthma exacerbation requiring oral corticosteroids or that required overnight hospitalisation requiring additional asthma treatment
* Uncontrolled disease or clinical abnormality
* Allergies to study drugs or the excipients
* Taking another investigational medication or prohibited medication
* Night shift workers
* Current smokers or subjects with a smoking history of at least 10 pack years

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 612 (Actual)
Dates: Start 2010-08-20; Primary Completion 2011-10-01 (Actual); Study Completion 2011-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (58):
- United States (22):
  - GSK Investigational Site, Bell Gardens, California
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Newport Beach, California
  - GSK Investigational Site, Riverside, California
  - GSK Investigational Site, Roseville, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Normal, Illinois
  - GSK Investigational Site, River Forest, Illinois
  - GSK Investigational Site, Columbia, Maryland
  - GSK Investigational Site, Rolla, Missouri
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Lake Oswego, Oregon
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Orangeburg, South Carolina
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Sugar Land, Texas
  - GSK Investigational Site, Murray, Utah
- Germany (7):
  - GSK Investigational Site, Mannheim, Baden-Wurttemberg
  - GSK Investigational Site, Oranienburg, Brandenburg
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Gelnhausen, Hesse
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- Japan (10):
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Hiroshima
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Ishikawa
  - GSK Investigational Site, Kagawa
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Kyoto
  - GSK Investigational Site, Okinawa
  - GSK Investigational Site, Tokyo
- Poland (4):
  - GSK Investigational Site, Tarnów
  - GSK Investigational Site, Tczew
  - GSK Investigational Site, Wroclaw
  - GSK Investigational Site, Zawadzkie
- Romania (8):
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Cluj-Napoca
  - GSK Investigational Site, Craiova
  - GSK Investigational Site, Deva
  - GSK Investigational Site, Piteşti
  - GSK Investigational Site, Ploieşti
  - GSK Investigational Site, Suceava
  - GSK Investigational Site, Timișoara
- Ukraine (7):
  - GSK Investigational Site, Dnipropetrovsk
  - GSK Investigational Site, Ivano-Frankivsk
  - GSK Investigational Site, Kharkiv
  - GSK Investigational Site, Kiev
  - GSK Investigational Site, Kyiv
  - GSK Investigational Site, Simferopol
  - GSK Investigational Site, Zaporizhia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] O'Byrne PM, Jacques L, Goldfrad C, Kwon N, Perrio M, Yates LJ, Busse WW. Integrated safety and efficacy analysis of once-daily fluticasone furoate for the treatment of asthma. Respir Res. 2016 Nov 24;17(1):157. doi: 10.1186/s12931-016-0473-x. PMID 27881132
- [Derived] Gross AS, Goldfrad C, Hozawa S, James MH, Clifton CS, Sugiyama Y, Jacques L. Ethnic sensitivity assessment of fluticasone furoate/vilanterol in East Asian asthma patients from randomized double-blind multicentre Phase IIb/III trials. BMC Pulm Med. 2015 Dec 24;15:165. doi: 10.1186/s12890-015-0159-z. PMID 26704701
- [Derived] Bleecker ER, Lotvall J, O'Byrne PM, Woodcock A, Busse WW, Kerwin EM, Forth R, Medley HV, Nunn C, Jacques L, Bateman ED. Fluticasone furoate-vilanterol 100-25 mcg compared with fluticasone furoate 100 mcg in asthma: a randomized trial. J Allergy Clin Immunol Pract. 2014 Sep-Oct;2(5):553-61. doi: 10.1016/j.jaip.2014.02.010. Epub 2014 Apr 24. PMID 25213048
- [Derived] Svedsater H, Jacques L, Goldfrad C, Bleecker ER. Ease of use of the ELLIPTA dry powder inhaler: data from three randomised controlled trials in patients with asthma. NPJ Prim Care Respir Med. 2014 Jun 26;24:14019. doi: 10.1038/npjpcrm.2014.19. No abstract available. PMID 24966061
- [Derived] Svedsater H, Dale P, Garrill K, Walker R, Woepse MW. Qualitative assessment of attributes and ease of use of the ELLIPTA dry powder inhaler for delivery of maintenance therapy for asthma and COPD. BMC Pulm Med. 2013 Dec 7;13:72. doi: 10.1186/1471-2466-13-72. PMID 24314123
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 106827 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 106827 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 106827 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 106827 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 106827 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 106827 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 106827 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants meeting eligibility criteria at the Screening visit completed a 4-week Run-in Period for Baseline safety evaluations and measures of asthma status. Participants were then randomized to a 12-week Treatment Period. 1110 participants were screened, 610 were randomized, and 609 received >=1 dose of study treatment.
Groups:
- Current Anti-asthma Therapy at a Fixed Dose: Participants were instructed to continue using an approved fixed dose of an inhaled corticosteroid (ICS) for 4 weeks. Participants were provided albuterol/salbutamol inhalation aerosol to be used as rescue medication during the Run-in Period.
- Placebo: Participants (par.) received placebo once daily (OD) in the evening from the dry powder inhaler (DPI) for 12 weeks. Participants were provided albuterol/salbutamol inhalation aerosol to be used as rescue medication during the Treatment Period.
- FF 100 µg OD: Participants received Fluticasone Furoate (FF) 100 microgram (µg) inhalation powder OD in the evening from the DPI for 12 weeks. Participants were provided albuterol/salbutamol inhalation aerosol to be used as rescue medication during the Treatment Period.
- FF/VI 100/25 µg OD: Participants received FF/Vilanterol (VI) 100/25 µg inhalation powder OD in the evening from the DPI for 12 weeks. Participants were provided albuterol/salbutamol inhalation aerosol to be used as rescue medication during the Treatment Period.
Period: Overall Study
Arm/Group | Current Anti-asthma Therapy at a Fixed Dose | Placebo | FF 100 µg OD | FF/VI 100/25 µg OD
Started | 0 | 203 | 205 | 201
Completed | 0 | 151 | 185 | 179
Not Completed | 0 | 52 | 20 | 22
Not completed — Adverse Event | 0 | 1 | 0 | 2
Not completed — Lack of Efficacy | 0 | 32 | 6 | 7
Not completed — Protocol Violation | 0 | 7 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 1 | 2
Not completed — Physician Decision | 0 | 6 | 7 | 6
Not completed — Withdrawal by Subject | 0 | 6 | 6 | 3

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Participants received placebo once daily (OD) in the evening from the dry powder inhaler (DPI) for 12 weeks. Participants were provided albuterol/salbutamol inhalation aerosol to be used as rescue medication during the Treatment Period.
- Total: Total of all reporting groups
Arm/Group | Placebo | FF 100 µg OD | FF/VI 100/25 µg OD | Total
Number analyzed (Participants) | 203 | 205 | 201 | 609
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.1 (16.49) | 40.4 (16.78) | 40.7 (16.38) | 39.7 (16.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 111 | 126 | 116 | 353
  Male | 92 | 79 | 85 | 256
Race/Ethnicity, Customized [Number; unit: participants]
  African American/African Heritage | 14 | 16 | 13 | 43
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian - Japanese Heritage | 19 | 16 | 15 | 50
  Asian - South East Asian Heritage | 0 | 0 | 1 | 1
  White - Arabic/North African Heritage | 0 | 1 | 0 | 1
  White - White/Caucasian/European Heritage | 169 | 170 | 172 | 511
  Mixed Race | 1 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Clinic Visit Trough (Pre-bronchodilator and Pre-dose) Forced Expiratory Volume in One Second (FEV1) at Week 12
Description: Pulmonary function was measured by FEV1, defined as the maximal amount of air that can be forcefully exhaled in one second. Trough FEV1 is defined as the clinic visit (pre-bronchodilator and pre-dose) FEV1measurement taken at the clinic visit while still on-treatment. Pre-dose and pre-rescue albuterol/salbutamol trough FEV1 was measured electronically by spirometry in the evening at the Baseline through Week 12 clinic visits. The highest of 3 technically acceptable measurements was recorded. Baseline was the pre-dose value obtained at Visit 3. Change from Baseline was calculated as the Week 12 value minus the Baseline value. The analysis was performed using an Analysis of Covariance (ANCOVA) model with covariates of Baseline trough FEV1, region, sex, age, and treatment group. The last observation carried forward (LOCF) method was used to impute missing data, in which the last non-missing post-Baseline on-treatment measurement at scheduled clinic visits was used to impute the missing m
Time Frame: Baseline and Week 12
Population: Intent-to-Treat (ITT) Population: all participants randomized to treatment, who received at least one dose of the study medication. Only those participants with non-missing covariates and post-Baseline FEV1 data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | FF 100 µg OD | FF/VI 100/25 µg OD
Number analyzed (Participants) | 193 | 203 | 200
Liters | 0.196 (0.0310) | 0.332 (0.0302) | 0.368 (0.0304)
Statistical Analysis 1: Comparison: Placebo vs FF 100 µg OD; Test type: Superiority or Other; p = 0.002, ANCOVA; Median Difference (Final Values) = 0.136, 95% CI 2-sided [0.051 to 0.222]
Statistical Analysis 2: Comparison: Placebo vs FF/VI 100/25 µg OD; Test type: Superiority or Other; p < 0.001, ANCOVA; Median Difference (Final Values) = 0.172, 95% CI 2-sided [0.087 to 0.258]
Statistical Analysis 3: Comparison: FF 100 µg OD vs FF/VI 100/25 µg OD; Test type: Superiority or Other; p = 0.405, ANCOVA; Median Difference (Final Values) = 0.036, 95% CI 2-sided [-0.048 to 0.120]

2. Primary Outcome: Change From Baseline in Weighted Mean Serial FEV1 Over 0-24 Hours Post-dose at Week 12
Description: Pulmonary function was measured by FEV1, defined as the maximal amount of air that can be forcefully exhaled in one second. Serial FEV1 measurements were taken electronically by spirometry at the Baseline and Week 12 clinic visits. Weighted mean was calculated using the 24-hour serial FEV1 measurements that included the pre-dose assessment (within 30 minutes prior to dosing at Baseline and within 5 minutes prior to dosing at Week 12) and post-dose assessments after 5, 15, and 30 minutes and 1, 2, 3, 4, 5, 12, 16, 20, 23, and 24 hours. At each time point, the highest of 3 technically acceptable measurements was recorded. Baseline was the value obtained at Visit 3. Change from Baseline was calculated as the average Week 12 FEV1 value minus the Baseline value. The analysis was performed using an ANCOVA model with covariates of Baseline FEV1, region, sex, age, and treatment group.
Time Frame: Baseline and Week 12
Population: ITT Population. Weighted mean serial FEV1 was calculated for the subset of participants for whom serial FEV1 was performed at Week 12.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | FF 100 µg OD | FF/VI 100/25 µg OD
Number analyzed (Participants) | 95 | 106 | 108
Liters | 0.212 (0.0456) | 0.398 (0.0432) | 0.513 (0.0430)
Statistical Analysis 1: Comparison: Placebo vs FF 100 µg OD; Test type: Superiority or Other; p = 0.003, ANCOVA; Median Difference (Final Values) = 0.186, 95% CI 2-sided [0.062 to 0.310]
Statistical Analysis 2: Comparison: Placebo vs FF/VI 100/25 µg OD; Test type: Superiority or Other; p < 0.001, ANCOVA; Median Difference (Final Values) = 0.302, 95% CI 2-sided [0.178 to 0.426]
Statistical Analysis 3: Comparison: FF 100 µg OD vs FF/VI 100/25 µg OD; Test type: Superiority or Other; p = 0.060, ANCOVA; Mean Difference (Final Values) = 0.116, 95% CI 2-sided [-0.005 to 0.236]

3. Secondary Outcome: Mean Change From Baseline in the Percentage of Rescue-free 24-hour (hr) Periods During the 12-week Treatment Period
Description: The number of inhalations of rescue albuterol/salbutamol inhalation aerosol used during the day and night was recorded by the participants in a daily electronic diary (eDiary). A 24-hour (hr) period in which a participant's responses to both the morning and evening assessments indicated no use of rescue medication was considered to be rescue free. The Baseline value was derived from the last 7 days of the daily eDiary prior to the randomization of the participant. Change from Baseline was calculated as the averaged value during the 12-week Treatment Period minus the Baseline value. The analysis was performed using an ANCOVA model with covariates of Baseline, region, sex, age, and treatment group.
Time Frame: Baseline and Week 12
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percentage of rescue-free 24-hr periods
Arm/Group | Placebo | FF 100 µg OD | FF/VI 100/25 µg OD
Number analyzed (Participants) | 202 | 204 | 201
Percentage of rescue-free 24-hr periods | 17.8 (2.26) | 26.5 (2.25) | 37.1 (2.26)

4. Secondary Outcome: Change From Baseline in the Percentage of Symptom-free 24-hour (hr) Periods During the 12-week Treatment Period
Description: Asthma symptoms were recorded in a daily eDairy by the participants every day in the morning and evening before taking any rescue or study medication and before the peak expiratory flow measurement. A 24-hour (hr) period in which a participant's responses to both the morning and evening assessments indicated no symptoms was considered to be symptom free. The Baseline value was derived from the last 7 days of the daily eDiary prior to the randomization of the participant. Change from Baseline was calculated as the averaged value during the 12-week Treatment Period minus the Baseline value. The analysis was performed using an ANCOVA model with covariates of Baseline, region, sex, age, and treatment group.
Time Frame: Baseline and Week 12
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percentage of symptom-free 24-hr periods
Arm/Group | Placebo | FF 100 µg OD | FF/VI 100/25 µg OD
Number analyzed (Participants) | 202 | 204 | 201
Percentage of symptom-free 24-hr periods | 14.6 (2.15) | 20.4 (2.13) | 32.5 (2.14)

5. Secondary Outcome: Change From Baseline in the Total Asthma Quality of Life Questionnaire (AQLQ) (+12) Score at Week 12/Early Withdrawal
Description: The AQLQ is a disease-specific, self-administered quality of life questionnaire used to evaluate the impact of asthma treatments on the quality of life of asthma sufferers. The AQLQ for 12 years and older (AQLQ [+12]) is a modified version of the AQLQ for use in asthma patients between the age of 12 and 70. The AQLQ contains 32 items in 4 domains: activity limitation (11 items), symptoms (12 items), emotional function (5 items), and environmental stimuli (4 items). For the 32 items on the questionnaire, the response format consists of a seven-point scale, where a value of 1 indicates "total impairment" and a value of 7 indicates "no impairment." The AQLQ total score is defined as the average of the scores from all 32 questions; thus, the total score ranges from 1 (indicates "total impairment") to 7 (indicates "no impairment"). Baseline was the total score obtained at Visit 3. Change from Baseline was calculated as the total score at Week 12 minus the total score at Baseline.
Time Frame: Baseline and Week 12/Early Withdrawal
Population: ITT Population. Only those participants available at the specified time points were analyzed. The analysis was performed using an ANCOVA model with covariates of Baseline, region, sex, age, and treatment group.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | FF 100 µg OD | FF/VI 100/25 µg OD
Number analyzed (Participants) | 149 | 184 | 180
Score on a scale | 0.61 (0.061) | 0.76 (0.055) | 0.91 (0.055)

6. Secondary Outcome: Number of Participants Who Withdrew Due to Lack of Efficacy During the 12-week Treatment Period
Description: The number of participants whose primary reason for withdrawal was lack of efficacy was analyzed.
Time Frame: From the first dose of the study medication up to Week 12/Early Withdrawal
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Placebo | FF 100 µg OD | FF/VI 100/25 µg OD
Number analyzed (Participants) | 203 | 205 | 201
participants | 32 | 6 | 7

7. Secondary Outcome: Serial FEV1 Over 0-1 Hour Post-dose at Randomization
Description: Pulmonary function was measured by FEV1, defined as the maximal amount of air that can be forcefully exhaled in one second. Serial FEV1 measurements were taken electronically by spirometry at Randomization. Serial FEV1 measurements after 5, 15, and 30 minutes and 1 hour post-dose were assessed. At each time point, the highest of 3 technically acceptable measurements was recorded. The analysis was performed using a repeated measures model adjusted for baseline, region, sex, age, treatment group, and planned time points.
Time Frame: Randomization
Population: ITT Population. Serial FEV1 was calculated for the subset of participants for whom serial FEV1 was performed. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles). Different participants may have been analyzed for different parameters, so the overall number of participants analyzed
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | FF 100 µg OD | FF/VI 100/25 µg OD
Number analyzed (Participants) | 203 | 205 | 201
Liters
  5 Minutes, n=117, 112, 117 | 2.489 (0.0308) | 2.493 (0.0314) | 2.484 (0.0308)
  15 Minutes, n=118, 115, 117 | 2.491 (0.0336) | 2.529 (0.0342) | 2.566 (0.0336)
  30 Minutes, n=118, 116, 118 | 2.532 (0.0354) | 2.552 (0.0359) | 2.596 (0.0354)
  1 Hour, n=119, 116, 119 | 2.552 (0.0344) | 2.571 (0.0350) | 2.674 (0.0344)

8. Other Pre Specified Outcome: Clinic Visit 12-hour Post-dose FEV1 at Week 12
Description: Pulmonary function was measured by FEV1, defined as the maximal amount of air that can be forcefully exhaled in one second. 12-hour post-dose FEV1 measurements were taken electronically by spirometry at the Week 12 clinic visit. The highest of 3 technically acceptable measurements was recorded. The analysis was performed using an ANCOVA model with covariates of Baseline FEV1, region, sex, age, and treatment group.
Time Frame: Week 12
Population: ITT Population. 12-hour post-dose FEV1 was analyzed in the subset of participants for whom serial FEV1 at Week 12 was performed.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | FF 100 µg OD | FF/VI 100/25 µg OD
Number analyzed (Participants) | 93 | 104 | 108
Liters | 2.462 (0.0502) | 2.674 (0.0475) | 2.830 (0.0468)

9. Other Pre Specified Outcome: Weighted Mean Serial FEV1 Over 0-24 Hours Post-dose at Baseline
Description: Pulmonary function was measured by FEV1, defined as the maximal amount of air that can be forcefully exhaled in one second. Serial FEV1 measurements were taken electronically by spirometry at Baseline. Weighted mean was calculated using the 24-hour serial FEV1 measurements that included the pre-dose assessment (within 30 minutes prior to dosing) and post-dose assessments after 5, 15, and 30 minutes and 1, 2, 3, 4, 5, 12, 16, 20, 23, and 24 hours. At each time point, the highest of 3 technically acceptable measurements were recorded. Baseline was the value obtained at Visit 3.
Time Frame: Baseline
Population: ITT Population. Weighted mean serial FEV1 was calculated in the subset of participants for whom serial FEV1 was performed.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Placebo | FF 100 µg OD | FF/VI 100/25 µg OD
Number analyzed (Participants) | 119 | 116 | 119
Liters | 2.543 (0.8494) | 2.552 (0.7527) | 2.709 (0.8153)

10. Other Pre Specified Outcome: Weighted Mean Serial FEV1 Over 0-4 Hours Post-dose at Baseline and Week 12
Description: Pulmonary function was measured by FEV1, defined as the maximal amount of air that can be forcefully exhaled in one second. Serial FEV1 measurements were taken electronically by spirometry at the Baseline and Week 12 clinic visits. Weighted mean serial FEV1 over 0-4 hours was calculated using the serial FEV1 measurements that included the pre-dose assessment (within 30 minutes prior to dosing at Baseline and within 5 minutes prior to dosing at Week 12) and post-dose assessments after 5, 15, and 30 minutes and 1, 2, 3, and 4 hours. At each time point, the highest of 3 technically acceptable measurements were recorded. Baseline was the value obtained at Visit 3.
Time Frame: Baseline and Week 12
Population: ITT Population. Weighted mean serial FEV1 was calculated in the subset of participants for whom serial FEV1 at Week 12 was performed. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Placebo | FF 100 µg OD | FF/VI 100/25 µg OD
Number analyzed (Participants) | 120 | 115 | 119
Liters
  Baseline, n=120, 115, 119 | 2.563 (0.8194) | 2.522 (0.7479) | 2.693 (0.7626)
  Week 12, n=96, 105, 109 | 2.636 (0.8519) | 2.657 (0.7912) | 2.894 (0.8383)

11. Other Pre Specified Outcome: Number of Participants With Bronchodilator Effect
Description: Bronchodilator effect is defined as an increase of FEV1 (defined as the maximal amount of air that can be forcefully exhaled in one second) from Baseline of both 12% and 200 milliliters (mL) during 24 hours, which was evaluated using the serial FEV1 measurements at Baseline (Visit 3).
Time Frame: Baseline
Population: ITT Population. Only the subset of participants performing serial measurements were analyzed.
Measure: Number; unit: participants
Arm/Group | Placebo | FF 100 µg OD | FF/VI 100/25 µg OD
Number analyzed (Participants) | 120 | 116 | 120
participants | 73 [0 to 272.0] | 77 [0 to 270.0] | 97 [0 to 62.0]

12. Other Pre Specified Outcome: Mean Change From Baseline in Daily Morning (AM) Peak Expiratory Flow (PEF) Averaged Over the 12-week Treatment Period
Description: Peak Expiratory Flow (PEF) is defined as the maximum airflow during a forced expiration beginning with the lungs fully inflated. PEF was measured by the participants using a hand-held electronic peak flow meter each morning prior to the dose of study medication and any rescue albuterol/salbutamol inhalation aerosol use. Change from Baseline (defined as the last 7 days prior to randomization of the participants) was calculated as the value of the averaged daily AM PEF over the 12-week treatment period (at Week 12) minus the Baseline value. The analysis was performed using an ANCOVA model with covariates of Baseline, region, sex, age, and treatment group.
Time Frame: From Baseline up to Week 12
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Liters per minute
Arm/Group | Placebo | FF 100 µg OD | FF/VI 100/25 µg OD
Number analyzed (Participants) | 103 | 204 | 201
Liters per minute | -0.4 (2.42) | 18.3 (2.41) | 32.9 (2.42)

13. Other Pre Specified Outcome: Mean Change From Baseline in Daily Evening (PM) PEF Averaged Over the 12-week Treatment Period
Description: PEF is defined as the maximum airflow during a forced expiration beginning with the lungs fully inflated. PEF was measured by the participants using a hand-held electronic peak flow meter each evening prior to the dose of study medication and any rescue albuterol/salbutamol inhalation aerosol use. Change from Baseline (defined as the last 7 days prior to randomization of the participants) was calculated as the value of the averaged daily PM PEF over the 12-week treatment period (at Week 12) minus the Baseline value. The analysis was performed using an ANCOVA model with covariates of Baseline, region, sex, age, and treatment group.
Time Frame: From Baseline up to Week 12
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Liters per minute
Arm/Group | Placebo | FF 100 µg OD | FF/VI 100/25 µg OD
Number analyzed (Participants) | 202 | 204 | 201
Liters per minute | -1.8 (2.36) | 14.1 (2.34) | 26.4 (2.35)

14. Other Pre Specified Outcome: Change From Baseline in the Asthma Control Test (ACT) Score at Week 12
Description: The ACT is a 5-item questionnaire developed as a measure of the participant's asthma control. Questions are designed to be self-completed by the participant and include the following: In the past 4 weeks, "How much of the time did your asthma keep you from getting as much done at work, school or at home?", "How often have you had shortness of breath?", "How often did your asthma symptoms wake you up at night or earlier than usual in the morning?", "How often have you used your rescue inhaler or nebulizer medication (such as albuterol)?" and "How would you rate your asthma control"? The ACT total score is defined as the sum of the scores from all 5 questions, provided all questions have been answered; thus, the total score ranges from 5 (poor control of asthma) to 25 (complete control of asthma). A score of 20 or higher indicates well-controlled asthma. Change from Baseline was calculated as the total score at Week 12/Early Withdrawal minus the total score at Baseline.
Time Frame: Baseline and Week 12/Early Withdrawal
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | FF 100 µg OD | FF/VI 100/25 µg OD
Number analyzed (Participants) | 154 | 189 | 185
Scores on a scale | 2.5 (0.26) | 3.8 (0.23) | 4.4 (0.23)

15. Other Pre Specified Outcome: Number of Participants With the Indicated Global Assessment of Change Responses at Week 4, Week 8, and Week 12/Early Withdrawal
Description: At the end of Week 4, Week 8, and Week 12/Early Withdrawal, the Global Assessment of Change Questionnaire that assesses changes in asthma symptoms (AS) and rescue medication use (RMU) was completed by the participants. The number of participants who chose the following answers to the questionnaire were determined: much better, somewhat better, a little better, the same, a little worse, somewhat worse, much worse (to assess the changes in asthma symptom); much less often , somewhat less often , a little less often , the same , a little more often , somewhat more often , much more often (to assess the changes in the frequency of rescue medication use).
Time Frame: Week 4, Week 8, and Week 12/Early Withdrawal
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Number; unit: participants
Arm/Group | Placebo | FF 100 µg OD | FF/VI 100/25 µg OD
Number analyzed (Participants) | 174 | 198 | 191
participants
  Week 4, AS - Much better, n=174, 198, 191 | 34 | 47 | 65
  Week 4, AS - Somewhat better, n=174, 198, 191 | 45 | 65 | 61
  Week 4, AS - A little better, n=174, 198, 191 | 42 | 47 | 37
  Week 4, AS - The same, n=174, 198, 191 | 33 | 29 | 23
  Week 4, AS - A little worse, n=174, 198, 191 | 6 | 10 | 3
  Week 4, AS - Somewhat worse, n=174, 198, 191 | 8 | 0 | 2
  Week 4, AS - Much worse, n=174, 198, 191 | 6 | 0 | 0
  Week 4, RMU - Much less often, n=174, 198, 191 | 39 | 59 | 75
  Week 4, RMU - Somewhat less often, n=174, 198, 191 | 40 | 48 | 51
  Week 4, RMU - A little less often, n=174, 198, 191 | 35 | 49 | 32
  Week 4, RMU - The same, n=174, 198, 191 | 31 | 33 | 28
  Week 4, RMU - A little more often, n=174, 198, 191 | 13 | 6 | 4
  Week 4, RMU - Somewhat more often, n=174, 198, 191 | 11 | 3 | 1
  Week 4, RMU - Much more often, n=174, 198, 191 | 5 | 0 | 0
  Week 8, AS - Much better, n=159, 192, 184 | 36 | 54 | 69
  Week 8, AS - Somewhat better, n=159, 192, 184 | 44 | 60 | 63
  Week 8, AS - A little better, n=159, 192, 184 | 38 | 40 | 22
  Week 8, AS - The same, n=159, 192, 184 | 29 | 33 | 24
  Week 8, AS - A little worse, n=159, 192, 184 | 7 | 5 | 3
  Week 8, AS - Somewhat worse, n=159, 192, 184 | 4 | 0 | 2
  Week 8, AS - Much worse, n=159, 192, 184 | 1 | 0 | 1
  Week 8, RMU - Much less often, n=159, 191, 184 | 37 | 65 | 86
  Week 8, RMU - Somewhat less often, n=159, 191, 184 | 32 | 48 | 43
  Week 8, RMU - A little less often, n=159, 191, 184 | 37 | 34 | 25
  Week 8, RMU - The same, n=159, 191, 184 | 36 | 39 | 23
  Week 8, RMU - A little more often, n=159, 191, 184 | 12 | 1 | 5
  Week 8, RMU - Somewhat more often, n=159, 191, 184 | 4 | 4 | 0
  Week 8, RMU - Much more often, n=159, 191, 184 | 1 | 0 | 2
  Week 12, AS - Much better, n=152, 187, 182 | 38 | 66 | 86
  Week 12, AS - Somewhat better, n=152, 187, 182 | 37 | 49 | 52
  Week 12, AS - A little better, n=152, 187, 182 | 29 | 35 | 13
  Week 12, AS - The same, n=152, 187, 182 | 29 | 30 | 23
  Week 12, AS - A little worse, n=152, 187, 182 | 9 | 7 | 7
  Week 12, AS - Somewhat worse, n=152, 187, 182 | 6 | 0 | 1
  Week 12, AS - Much worse, n=152, 187, 182 | 4 | 0 | 0
  Week 12, RMU - Much less often, n=150, 187, 182 | 42 | 76 | 89
  Week 12, RMU -Somewhat less often, n=150, 187, 182 | 32 | 46 | 43
  Week 12, RMU -A little less often, n=150, 187, 182 | 24 | 25 | 21
  Week 12, RMU - The same, n=150, 187, 182 | 34 | 32 | 23
  Week 12, RMU -A little more often, n=150, 187, 182 | 12 | 6 | 5
  Week 12, RMU -Somewhat more often, n=150, 187, 182 | 3 | 1 | 1
  Week 12, RMU - Much more often, n=150, 187, 182 | 3 | 1 | 0

16. Other Pre Specified Outcome: Number of the Indicated Unscheduled Asthma-related Healthcare Visits During the Treatment Period
Description: All unscheduled asthma-related visits to a physician's office, visits to urgent care, visits to the emergency department, and hospitalizations (ICU=intensive care unit; GW=general ward) associated with severe asthma exacerbations or other asthma-related healthcare were recorded.
Time Frame: From Baseline up to Week 12/Early Withdrawal
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Number of visits
Arm/Group | Placebo | FF 100 µg OD | FF/VI 100/25 µg OD
Number analyzed (Participants) | 203 | 205 | 201
Number of visits
  Number of Home Visits (Day) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)
  Number of Home Visits (Night) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)
  Number of Physician Office/Practice Visits | 0.0 (0.24) | 0.0 (0.39) | 0.0 (0.10)
  Number of Urgent Care/Outpatient Clinic Visits | 0.0 (0.07) | 0.0 (0.07) | 0.0 (0.00)
  Number of Emergency Room Visits | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)
  Number of Inpatient Hospitalization Days (ICU) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)
  Number of Inpatient Hospitalization (GW) Days | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)

17. Other Pre Specified Outcome: Number of Participants Who Used the Inhaler Correctly or Incorrectly at Baseline, Week 2, and Week 4
Description: Participants were given a demonstration of correct inhaler use (using placebo inhalers), and the participants' competence to correctly use the demonstration inhaler was then assessed.
Time Frame: Baseline (BL), Week 2 (W2), and Week 4 (W4)
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Number; unit: participants
Arm/Group | Placebo | FF 100 µg OD | FF/VI 100/25 µg OD
Number analyzed (Participants) | 203 | 205 | 201
participants
  BL: Used Inhaler Correctly, n=203, 205, 201 | 194 | 196 | 188
  BL: Used Inhaler Incorrectly, n=203, 205, 201 | 9 | 9 | 13
  W2: Used Inhaler Correctly, n=190, 203, 200 | 190 | 203 | 200
  W2: Used Inhaler Incorrectly, n=190, 203, 200 | 0 | 0 | 0
  W4: Used Inhaler Correctly, n=175, 199, 195 | 175 | 199 | 195
  W4: Used Inhaler Incorrectly, n=175, 199, 195 | 0 | 0 | 0

18. Other Pre Specified Outcome: Number of Participants With the Indicated Reason for Incorrect Inhaler Use and Who Required Additional Instruction the Indicated Number of Times at Baseline, Week 2, and Week 4
Description: Participants were given a demonstration of correct inhaler use (using placebo inhalers), and the participants' competence to correctly use the demonstration inhaler was then assessed based on 3 steps: open the device, inhale the dose, and close the device. If the participants did not perform the maneuvers correctly, the step of the inhaler use that was performed incorrectly by the participants was recorded. The entire procedure was demonstrated once again. and the number of times that the participants required additional instruction (RAI) was recorded.
Time Frame: Baseline, Week 2, and Week 4
Population: ITT Population. Only those participants who used the inhaler incorrectly at the specified time points were analyzed.
Measure: Number; unit: participants
Arm/Group | Placebo | FF 100 µg OD | FF/VI 100/25 µg OD
Number analyzed (Participants) | 9 | 9 | 13
participants
  BL: Opened the Device Incorrectly, n= 9, 9, 13 | 8 | 4 | 6
  BL: Inhaled the Dose Incorrectly, n= 9, 9, 13 | 1 | 5 | 6
  BL: Closed the Device Incorrectly, n= 9, 9, 13 | 1 | 0 | 1
  BL: RAI once, n= 9, 9, 13 | 9 | 5 | 8
  BL: RAI 2 Times, n= 9, 9, 13 | 0 | 4 | 4
  BL: RAI 3 Times, n= 9, 9, 13 | 0 | 0 | 1
  BL: RAI >3 Times, n= 9, 9, 13 | 0 | 0 | 0
  W2: Opened the Device Incorrectly, n= 0, 0, 0 | NA — No participants used the inhaler incorrectly at Week 2; thus, no data can be reported at this time point. | NA — No participants used the inhaler incorrectly at Week 2; thus, no data can be reported at this time point. | NA — No participants used the inhaler incorrectly at Week 2; thus, no data can be reported at this time point.
  W2: Inhaled the Dose Incorrectly, n= 0, 0, 0 | NA — No participants used the inhaler incorrectly at Week 2; thus, no data can be reported at this time point. | NA — No participants used the inhaler incorrectly at Week 2; thus, no data can be reported at this time point. | NA — No participants used the inhaler incorrectly at Week 2; thus, no data can be reported at this time point.
  W2: Closed the Device Incorrectly, n= 0, 0, 0 | NA — No participants used the inhaler incorrectly at Week 2; thus, no data can be reported at this time point. | NA — No participants used the inhaler incorrectly at Week 2; thus, no data can be reported at this time point. | NA — No participants used the inhaler incorrectly at Week 2; thus, no data can be reported at this time point.
  W2: RAI once, n= 0, 0, 0 | NA — No participants used the inhaler incorrectly at Week 2; thus, no participants required additional instruction. | NA — No participants used the inhaler incorrectly at Week 2; thus, no participants required additional instruction. | NA — No participants used the inhaler incorrectly at Week 2; thus, no participants required additional instruction.
  W2: RAI 2 Times, n= 0, 0, 0, | NA — No participants used the inhaler incorrectly at Week 2; thus, no participants required additional instruction. | NA — No participants used the inhaler incorrectly at Week 2; thus, no participants required additional instruction. | NA — No participants used the inhaler incorrectly at Week 2; thus, no participants required additional instruction.
  W2: RAI 3 Times, n= 0, 0, 0 | NA — No participants used the inhaler incorrectly at Week 2; thus, no participants required additional instruction. | NA — No participants used the inhaler incorrectly at Week 2; thus, no participants required additional instruction. | NA — No participants used the inhaler incorrectly at Week 2; thus, no participants required additional instruction.
  W4: Opened the Device Incorrectly, n= 0, 0, 0 | NA — No participants used the inhaler incorrectly at Week 4; thus, no data can be reported at this time point. | NA — No participants used the inhaler incorrectly at Week 4; thus, no data can be reported at this time point. | NA — No participants used the inhaler incorrectly at Week 4; thus, no data can be reported at this time point.
  W4: Inhaled the Dose Incorrectly, n= 0, 0, 0 | NA — No participants used the inhaler incorrectly at Week 4; thus, no data can be reported at this time point. | NA — No participants used the inhaler incorrectly at Week 4; thus, no data can be reported at this time point. | NA — No participants used the inhaler incorrectly at Week 4; thus, no data can be reported at this time point.
  W4: Closed the Device Incorrectly, n= 0, 0, 0 | NA — No participants used the inhaler incorrectly at Week 4; thus, no data can be reported at this time point. | NA — No participants used the inhaler incorrectly at Week 4; thus, no data can be reported at this time point. | NA — No participants used the inhaler incorrectly at Week 4; thus, no data can be reported at this time point.
  W4: RAI once, n= 0, 0, 0 | NA — No participants used the inhaler incorrectly at Week 4; thus, no participants required additional instruction. | NA — No participants used the inhaler incorrectly at Week 4; thus, no participants required additional instruction. | NA — No participants used the inhaler incorrectly at Week 4; thus, no participants required additional instruction.
  W4: RAI 2 Times, n= 0, 0, 0 | NA — No participants used the inhaler incorrectly at Week 4; thus, no participants required additional instruction. | NA — No participants used the inhaler incorrectly at Week 4; thus, no participants required additional instruction. | NA — No participants used the inhaler incorrectly at Week 4; thus, no participants required additional instruction.
  W4: RAI 3 Times, n= 0, 0, 0 | NA — No participants used the inhaler incorrectly at Week 4; thus, no participants required additional instruction. | NA — No participants used the inhaler incorrectly at Week 4; thus, no participants required additional instruction. | NA — No participants used the inhaler incorrectly at Week 4; thus, no participants required additional instruction.
  W4: RAI >3 Times, n= 0, 0, 0 | NA — No participants used the inhaler incorrectly at Week 4; thus, no participants required additional instruction. | NA — No participants used the inhaler incorrectly at Week 4; thus, no participants required additional instruction. | NA — No participants used the inhaler incorrectly at Week 4; thus, no participants required additional instruction.

ADVERSE EVENTS:
Time Frame: Serious Adverse Events (SAEs) and non-serious AEs were collected from the first dose of study medication up to Week 12/Early Withdrawal.
Description: SAEs and AEs were collected in members of Intent-to-Treat (ITT) Population, comprised of all participants randomized to treatment, who received at least one dose of the study medication.
Arm/Group | Placebo | FF 100 µg OD | FF/VI 100/25 µg OD
Serious Adverse Events (participants affected / at risk) | 0/203 | 1/205 | 0/201
Other Adverse Events (participants affected / at risk) | 22/203 | 20/205 | 29/201
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=203) | FF 100 µg OD (N=205) | FF/VI 100/25 µg OD (N=201)
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=203) | FF 100 µg OD (N=205) | FF/VI 100/25 µg OD (N=201)
Nasopharyngitis (Infections and infestations) | 15 | 14 | 20
Headache (Nervous system disorders) | 8 | 9 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.